CLINICAL TRIAL: NCT00836940
Title: A 12-week Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Evaluate Safety, Tolerability, and Efficacy of GRC 8200, a New Oral DPP -IV Inhibitor, in Patients With Type 2 Diabetes Mellitus.
Brief Title: A Clinical Study of GRC 8200 in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glenmark Pharmaceuticals Europe Ltd. (R&D) (Industry)
Responsible Party: Dr Manmath Patekar, Glenmark Pharmaceuticals ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GRC 8200-301
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; GRC 8200
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Placebo Comparator)
  Interventions: Drug: GRC 8200
- 2 (Experimental): GRC 8200-25mg OD
  Interventions: Drug: GRC 8200
- 3 (Experimental): GRC 8200-50mg OD
  Interventions: Drug: GRC 8200
- 4 (Experimental): GRC 8200-50mg BD
  Interventions: Drug: GRC 8200
- 5 (Experimental): GRC 8200-100mg OD
  Interventions: Drug: GRC 8200

INTERVENTIONS:
Drug: GRC 8200 — Capsules, 25 to 100mg, once/ twice a day, 12 weeks

SUMMARY:
The study is aimed at evaluating efficacy and safety of GRC 8200 in type 2 diabetes mellitus patients.

The study involves six weeks of wash out period and two weeks run in period for patients currently on mono-therapy and a two week run in period only for drug naïve patients.

This is a placebo controlled study. One of the five treatment arms is placebo. The duration of treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥30 years of age
* At screening, females of non-childbearing potential or females of childbearing potential with adequate contraception
* Has an established clinical diagnosis of type 2 diabetes mellitus for at least 3 months prior to the screening period
* Is being treated for diabetes either with diet and exercise alone, or on monotherapy with any of the antidiabetic drugs
* Has an HbA1c value at screening between 6.5% and 10%

Exclusion Criteria:

* Has type 1 diabetes
* Is a female who is lactating or is pregnant
* Has a history of acute metabolic diabetic complications
* Has clinically significant disease other than type 2 diabetes mellitus

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c compared with placebo at the end of 12 week treatment period | 12 weeks

SECONDARY OUTCOMES:
Change in HbA1c from baseline at the end of 4 and 8 weeks of treatment | 4 and 8 weeks
Fasting plasma glucose and fasting serum insulin | 12 weeks
Plasma glucose 2 hours post glucose challenge (OGTT) | 12 weeks
HOMA-IR | 12 weeks
HOMA-B | 12 weeks
Change in serum lipids | 12 weeks
Body weight | 12 weeks
Waist circumference | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Glenmark Investigational site, Mumbai, India